CLINICAL TRIAL: NCT06405204
Title: The Effect of Myo-inositol, Melatonin and Co-enzyme q10 on Ovarian Reserve Parameters and Intra-cytoplasmic Sperm Injection Outcomes in Patient With Poor Ovarian Reserve: an Open Label Randomized Clinical Trial
Brief Title: of Myo-inositol, Melatonin and Co-enzyme q10 on Ovarian Reserve
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Co-enzyme q10
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: IVF
Keywords: Myo-inositol; Melatonin; Co-enzyme q10; ovarian reserve
MeSH Terms: interventions — Inositol; coenzyme Q10; Melatonin; Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- myo-inositol (Experimental): myo-inositol (1gm capsules bd ) plus folic acid 400 mcg per day
  Interventions: Drug: Myoinositol
- melatonin (Experimental): melatonin 1 capsule every night orally before going to bed plus folic acid 400mcg per day
  Interventions: Drug: Melatonin
- co-enzyme Q10 (Experimental): co-enzyme Q10 100mg per day plus folic acid 400 mcg per day
  Interventions: Drug: Co-Enzyme Q10
- control group. (Placebo Comparator): will receive folic acid 400 mcg per day
  Interventions: Drug: Folic acid

INTERVENTIONS:
Drug: Myoinositol — an enzymatic isoform of inositol and belongs to the vitamin B complex family
  Other Names: femtonex; Viocyst
  Arms: myo-inositol
Drug: Co-Enzyme Q10 — a lipid-soluble quinone, acting as an effective antioxidant,
  Other Names: Co Q
  Arms: co-enzyme Q10
Drug: Melatonin — an indoleamine with low molecular weight that is synthesized by different cells and organs in the body. More importantly, melatonin is an outstanding antioxidant
  Arms: melatonin
Drug: Folic acid — control
  Other Names: folicap
  Arms: control group.

SUMMARY:
To evaluate the role of Myo-inositol, melatonin and co-enzyme Q10 on ovarian reserve parameters and ICSI outcome in poor ovarian responder

DETAILED DESCRIPTION:
Each patient will be subjected to:

Full history taking. Systematic clinical examination to assess the general condition, body mass index (BMI) and local pelvic physical findings and AFC by trans-vaginal ultrasound on day 2 to day 3 of menstruation. Routine labs as CBC, liver & kidney functions to exclude general disease as a contraindication for induction or pregnancy.

Blood sample will be obtained for assessment of basal serum levels of FSH, LH, E2 on days 2- 3 of the cycle. PRL, AMH and TSH Ovarian Stimulation The patients will begin injections of recombinant FSH (rFSH, Gonal-F; Merck- Serono, Italy) from day 2-3 of menstruation, with daily dose of 300-450 IU adjusted according to individual conditions on the basis of the antral follicle count (AFC),hormonal profile, age, body mass index (BMI), and previous ovarian response, according to the standard operating procedures of the center. . For pituitary suppression, the patients will receive GnRH antagonist Cetrorelix (CETROTIDE 0.25Mg/d, Merck Serono, Germany) 0.25 mg/day subcutaneously from day 6 of induction until trigger day. The serum LH, estradiol levels as well as number and size of follicles will be monitored every two days, starting from stimulation day 6 until the day of hCG injection

ELIGIBILITY:
Inclusion Criteria:

* Infertile women who have one of the criteria of poor ovarian response as follows;

  * Antral follicle count less than 7
  * Anti-Mullerian hormone level Less than 1.2 ng/ml

Exclusion Criteria:

1. Any endocrine or metabolic disorder such as hyperprolactinemia, diabetes and thyroid dysfunction
2. Any pelvic pathology such as hydrosalpinx, uterine anomaly.
3. Any male factor infertility such as Oligo-Astheno-Teratozoospermia (OAT) or azoospermia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 1 month of induction for ICSI trial
  serum HCG positive

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Salem, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No